CLINICAL TRIAL: NCT01049256
Title: Developing an Improved Measure of Chemosensitivity for the Study of Periodic Breathing in Heart Failure: the Cyclocapnic Method
Brief Title: The Cyclocapnic Method for Measurement of Chemosensitivity
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Darrel Francis, Imperial College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07/H0712/129
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Periodic Breathing; Heart Failure
Keywords: Periodic breathing; Heart Failure; Chemoreflex; Chemosensitivity
MeSH Terms: conditions — Heart Failure | interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: carbon dioxide — sinusoidal carbon dioxide administration

SUMMARY:
We aim to test our method for measuring chemosensitivity (the ventilatory response to a change in carbon dioxide), which uses sinusoidal carbon dioxide stimuli.

Hypotheses:

* Carbon dioxide sensitivity is dependent on the cycle time over which we administer the gas (frequency).
* Chemoreflex gain decreases as deadspace increases.

DETAILED DESCRIPTION:
We will apply a new method for the measurement of chemosensitivity (how sensitive a person is to changes in carbon dioxide), which is one of the principle determinants of whether people with heart failure develop abnormal breathing patterns We have shown in a pilot study that administering sinusoidal patterns of inspired carbon dioxide produces similar sinusoidal responses in ventilation. We aim to test our method for measuring chemosensitivity, which uses sinusoidal carbon dioxide stimuli (similar to those that drive the oscillations in ventilation found in periodic breathing). We aim to show that how the cycle time of carbon dioxide administered affects the resulting ventilatory oscillations and therefore that when measuring the chemoreflex clinically, it is important to deliver carbon dioxide stimuli that replicate the cycle time of oscillations in carbon dioxide seen in periodic breathing (typically approximately one minute).

ELIGIBILITY:
Inclusion Criteria:

* Heart failure subjects with stable cardiorespiratory control to be recruited from our institution's specialist heart failure clinic.
* Normal healthy volunteers, with normal systolic function.

Exclusion Criteria:

* We will exclude patients with chronic respiratory disease (every patient will have formal lung function testing on entrance into the study) or unstable coronary artery disease (myocardial infarction or unstable angina within the past 3 months).
* In addition any subjects receiving treatment with morphine and derivatives, theophylline, oxygen, benzodiazepines or acetazolamide will be excluded as these affect chemosensitivity.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Chemoreflex gain as measured by cyclocapnic method | every minute

CONTACTS AND LOCATIONS:
Overall Officials: Darrel P Francis, MD, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, London, United Kingdom